CLINICAL TRIAL: NCT06573658
Title: Short-term Neurophysiological Changes After a Perturbation-based Training in Community-dwelling Older Adults: A Pilot Study
Brief Title: Neurophysiological Changes After Perturbation-based Training in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20230928002
Record Dates: First submitted 2024-07-30; First posted 2024-08-27 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Falling; Community Dwelling Older Adults; Postural Stability; Brain Connectivity; Brain Structure
Keywords: Perturbation; Magnetic Resonance Image; MRI; step training; responsive postural control; balance; external disturbance; fall

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to PBT or active control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perturbation-based balance training group (Experimental): This group will receive two sessions of treadmill walking at their comfortable speed involving perturbations
  Interventions: Behavioral: Perturbation-based balance training (PBT)
- Control (Placebo Comparator): This group will receive two sessions of treadmill walking at their comfortable speed involving no perturbations
  Interventions: Behavioral: Walking exercise (control)

INTERVENTIONS:
Behavioral: Perturbation-based balance training (PBT) — It will be a two-session training with each session lasting for approximately an hour. Perturbations will be induced during treadmill walking. Participants will be instructed to recover their balance and continue walking after the perturbations.
  Arms: Perturbation-based balance training group
Behavioral: Walking exercise (control) — It will be a two-session training with each session lasting for approximately an hour. The same training duration and format will be used as the PBT group, except that no perturbations will be induced during the treadmill walking.
  Arms: Control

SUMMARY:
This is an assessor-blinded neurophysiological study. Participants will be randomly assigned to a perturbation-based training (PBT) or a walking (control) group. Changes in postural stability and neurophysiology in the brain following PBT compared to walking exercise without perturbation will be investigated.

DETAILED DESCRIPTION:
A total of 88 participants will be randomly assigned to two groups receiving perturbation-based training (PBT) or walking exercise without perturbation (control). Written informed consent will be obtained from participants prior to the baseline assessment. The study will be reported and conducted in line with the CONSORT statement. Participants will be recruited via convenience sampling in the local community. Both groups will receive two sessions of treadmill walking at their comfortable speed. Perturbations will be induced during treadmill walking only for the PBT group. As informed from previous literature, two sessions of PBT could have improved postural stability for up to 1.5 years. Between-group differences in behavioural and MRI findings will be examined before and after training to identify training-induced changes in postural stability, brain structures, and functional connectivities. Retention of the changes in the postural stability will be assessed four months after the training period. Incidents of falls will be followed up for 12 months after training.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 60 years old
* Community-dwelling
* Right-handed
* Able to communicate effectively in Cantonese or Mandarin
* Able to walk independently on level ground for ≥ 30 minutes
* Abbreviated Mental Test (Hong Kong version) score ≥ 6

Exclusion Criteria:

* Metal implants (e.g. pacemaker, artificial cochlea)
* Uncorrected vision or hearing impairment
* Osteoporosis
* Hip or knee replacement within the last year
* Musculoskeletal, cardiovascular, mental, or neurological disorders (such as Parkinson's disease) which can affect MRI examination, balance control, or exercise participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Gray matter density in arbitrary units by structural Magnetic Resonance Imaging | pre-intervention, and within 1-week after the intervention
  Gray matter density at cortical and subcortical regions will be taken by structural MRI. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.
Brain connectivity derived from the correlation between the Blood-oxygen-level-dependent (BOLD) signals from different brain regions in arbitrary units obtained during functional MRI | pre-intervention, and within 1-week after the intervention
  BOLD signal reflecting the brain connectivity during rest will be taken through resting-state functional MRI, during which subjects are instructed to relax with eyes open, to let their mind wander, and not think of anything specific. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.

SECONDARY OUTCOMES:
Postural stability | pre-intervention, within 1 week after intervention and 4 months after intervention
  Postural stability at the recovery steps after the perturbation will be calculated as the distance between the absolute CoM position in an anteroposterior direction relative to the closest edge of Base of Support (BoS) and normalized by foot length.
  The absolute CoM position and BoS position will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.
Number of laboratory-falls | pre-intervention, within 1 week after intervention and 4 months after intervention
  The number of laboratory-falls following perturbation during assessment sessions will be recorded. A fall will be defined if there is a body-weight support of 30% or more from the full-body safety harness.
Number of real-life-falls | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 7 months, 8 months, 9 months, 10 months, 11 months, and 12 months after the intervention.
  The number of real-life falls in 12 months after randomization will be recorded. Fall circumstances and related injuries will be enquired via phone contact. A fall is defined as an event resulting in a person unintentionally coming to rest on the ground or other lower level, not as the result of a major intrinsic event e.g., syncope, stroke, seizure, or overwhelming hazard such as an earthquake.
Step time of the recovery steps in milliseconds (ms) | pre-intervention, within 1 week after intervention and 4 months after intervention
  Step time of the recovery steps after the perturbation will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.
Step length of the recovery steps in millimeters (mm) | pre-intervention, within 1 week after intervention and 4 months after intervention
  Step length of the recovery steps after the perturbation will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.
Trunk angle | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention
  The trunk angle at the recovery steps after the perturbation will be calculated as the angle between the trunk segment with the vertical line. The position of the trunk will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.
Hip height in millimeters (mm) | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention
  Hip height at the recovery steps after the perturbation will be calculated as the vertical distance from the ground to the midpoint of bilateral hips and normalized by the subjects' height. The positions of bilateral hips will be traced by the motion capture system synchronized with the force plates embedded underneath the slip-treadmill belts.
Responsive postural adjustment upon translation | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention
  Responsive postural adjustment upon translation will be assessed through Motor Control Test on a computerized dynamic posturography (Bertec® Balance Advantage® Dynamic System, Bertec® Corporation, Columbus, USA). During the Motor Control Test, participants will be requested to maintain their standing balance in response to 18 translations of the standing platform in either forward or backward direction with small, medium or large amplitudes. Weight symmetry, latency of reaction, and amplitude of sway will be recorded. Full-body safety harness will be worn throughout the tests to protect the participants from any potential loss of balance.
Responsive postural adjustment upon tilting | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention
  Responsive postural adjustment upon tilting will be assessed through Adaptation Test on a computerized dynamic posturography (Bertec® Balance Advantage® Dynamic System, Bertec® Corporation, Columbus, USA). During the Adaptation Test, the force platform will either tilt up or down for a total of 10 repetitions. Sway energy will be recorded. Full-body safety harness will be worn throughout the tests to protect the participants from any potential loss of balance.
Muscle activation onset latency in milliseconds | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention
  Muscle latency will be collected from trunk and leg muscles using electromyography.
Balance confidence | pre-intervention, immediately after the intervention, 1 week after intervention and 4 months after intervention, and at the last prospective fall follow-up
  Balance confidence will be measured with the Chinese version of the shortened version of Activities-Specific Balance Confidence Scale (ABC-6). The scale value is from 0 to 100, with higher values representing higher balance confidence.
Cognitive flexibility and executive function | pre-intervention, immediately after the intervention, 1 week after intervention, and 4 months after intervention
  Cognitive flexibility and executive function assessed by Trial Making Tests A and B (in the unit of seconds)
Functional lower body strength | pre-intervention, immediately after the intervention, 1 week after intervention, and 4 months after intervention
  Functional lower body strength will be assessed by Five-time Sit to Stand Test (in the unit of seconds)
Dynamic balance | pre-intervention, immediately after the intervention, 1 week after intervention, and 4 months after intervention
  Dynamic balance will be assessed by Alternate Step Test (in the unit of seconds)
Mobility | pre-intervention, immediately after the intervention, 1 week after intervention, and 4 months after intervention
  Mobility will be assessed by Timed Up and Go test (in the unit of seconds).
White matter density in arbitrary units by structural Magnetic Resonance Imaging | pre-intervention, and immediately after the intervention
  White matter density at cortical and subcortical regions will be taken by structural MRI. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.
Gray matter volume in cubic millimeters (mm³) by structural Magnetic Resonance Imaging (MRI) | pre-intervention, and immediately after the intervention
  Gray matter volume at cortical and subcortical regions will be measured by Structural MRI. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.
White matter volume in cubic millimeters (mm³) by structural Magnetic Resonance Imaging (MRI) | pre-intervention, and immediately after the intervention
  White matter volume at cortical and subcortical regions will be measured by Structural MRI. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.
Cortical thickness in mm measured by structural Magnetic Resonance Imaging | pre-intervention, and immediately after the intervention
  Cortical thickness in mm measured by structural MRI. The regions of interest include the cerebellar, inferior parietal, occipital, and frontal cortices.
Fractional anisotropy ranges from 0-1 derived from Diffusion Tensor Imaging | pre-intervention, and immediately after the intervention
  The degree of anisotropy of water diffusion in white matter tracts will be derived from the diffusion tensor. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.
Mean diffusivity measures in mm²/s by Diffusion Tensor Imaging | pre-intervention, and immediately after the intervention
  Mean diffusivity will be derived from the diffusion tensor. The regions of interest include the cerebellum, basal ganglia, thalamus, hippocampus, inferior parietal cortex, occipital and frontal lobe.

CONTACTS AND LOCATIONS:
Overall Officials: Sau Lan Tsang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No